CLINICAL TRIAL: NCT04384861
Title: Phase Three: Improving Physician Empathy, Compassionate Care and Wellness Through the Development of Resilience-building Communities of Practice and Creating a Culture of Empathy.
Brief Title: Improving Physician Empathy, Compassionate Care and Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Edward Spilg, Assistant Professor and Research Chair in Physician Wellness, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20180536-01H
Record Dates: First submitted 2020-04-28; First posted 2020-05-12 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Burnout, Professional; Resilience; Stress, Emotional
Keywords: Professional Burnout; Wellness; Emotional Stress; Resilience
MeSH Terms: conditions — Burnout, Professional; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Physician volunteers were first divided by gender and then randomly assigned to either the CONTROL (no SMART Wellness training) or ACTIVE (received SMART Wellness training) arms of the study.
Who Masked: Participant
Masking Description: Because the SMART training & Focus Groups were done in groups, ACTIVE participants were not masked from each other or the Investigators. Because the CONTROL participants did not attend any in-person meetings, they were masked from each other, the ACTIVE participants and the Investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTIVE (Experimental): The ACTIVE arm of the project received the Mayo Clinic SMART training (1 two-hour in-person workshop) and access to the Mayo Clinic's SMART eLearning Support study modules (4 x 45 minute modules in weeks 1-4; 20 x 10 minute modules weeks 5-24)
  Interventions: Behavioral: Mayo Clinic SMART program (Stress Management and Resilience Training)
- CONTROL (No Intervention): The CONTROL did not receive any interventions.

INTERVENTIONS:
Behavioral: Mayo Clinic SMART program (Stress Management and Resilience Training) — The SMART program included a workshop and ongoing eLearning Support. The learning objectives of the workshop are: (1) learn the neuroscience and behavioural aspects of human experience, particularly with respect to stress, resiliency, performance and wellness and (2) learn practical approaches to enhance engagement and emotional intelligence and thereby decrease stress and anxiety, increase resilience, enhance performance, and improve relationships. The goal of the eLearning support is to support and reinforce the messages and techniques delivered in the 2-hour workshop.
  Other Names: Mayo Clinic SMART eLearning Support
  Arms: ACTIVE

SUMMARY:
Background

Definitions of resilience vary according to the context in which it is discussed. It is often considered from the perspective of the individual. Connor & Davidsondescribe it as "the personal qualities that enable an individual to thrive in the face of adversity". Various studies have now shown a link between individual resilience and various mental health outcomes such as burnout, secondary traumatic stress, depression, and anxiety. In a systematic review by Fox et al., 22 studies explicitly stated an aim of improving physician resilience. However, there was a lack of consensus concerning the conceptual understanding of resilience with low methodological rigour of the included studies.

Research Questions

1. What effect will an evidence-based resilience building intervention have on levels of resilience, stress and subjective happiness in Department of Medicine Faculty at the University of Ottawa?
2. How might implementation of an evidence-based resilience building intervention on Department of Medicine faculty, lead to the development of a community of practice for physician wellness in the Department of Medicine at The Ottawa Hospital/University of Ottawa?

Methods All academic physicians in the Department of Medicine, University of Ottawa were invited to participate. We recruited 40 participants in total, randomized to either the ACTIVE or CONTROL groups.

Workshop ACTIVE participants (Group A) attended a 2-hour Stress Management and Resiliency Training (SMART) program developed by the Mayo Clinic. CONTROL (Group B) participants did not attend this training.

Questionnaires Both Group A & B completed questionnaires on resilience, perceived stress, anxiety and happiness at 0 weeks (pre-training) and 12 and 24-weeks post training.

E-learning support Following completion of the 2-hour workshop, Group A participants were enrolled in an online e-learning support program on a website developed by the Mayo Clinic. The aim of this was to support and reinforce the messages and techniques delivered in the 2-hour workshop. Participants were invited to participate for either 12 or 24 weeks.

Focus groups Group A participants were invited to join a focus group 12 weeks after the workshop was run. These focus groups explored themes of resilience, stress, and burnout.

Analysis of Results Quantitative (Questionnaires): For each measurement scale, the change from baseline will be compared between groups (Active Arm and Control Arm) using the two-sample t-test. To supplement these analyses, the within-group change (baseline vs week 4/12/24) will be assessed for the Active Arm using the paired t-test. A sample size of 40 was selected for this study after weighing statistical considerations along with logistical and resource constraints. In general, for a continuous outcome variable, a sample size of 40 provides statistical power (two-tailed, alpha=0.05) of >85% to detect a difference of 1 standard deviation between groups.

Qualitative (Focus Groups): Constructivist grounded theory informed the iterative data collection and analysis process. Transcripts were analysed using a three-staged process of initial, focused, and theoretical coding. Themes will be identified using constant comparative analysis and grouped to look at the interrelationship of categories.

ELIGIBILITY:
Inclusion Criteria:

* a full-time physician within the Department of Medicine at the Ottawa Hospital

Exclusion Criteria:

* part-time physicians; those external to the department

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Change in Connor-Davidson Resilience Scale (CD-RISC) scores | Administered prior to the intervention, and then at 12 and 24 weeks post-intervention
  * utilized for the assessment of the self-reported measures of resilience and the ability to cope with adversity
  * 25 questions; responses from 0 to 4
  * minimum total score: 0; maximum total score 100; higher scores indicative of greater levels of resilience.
Change in Perceived Stress Scale (PSS) scores | Administered prior to the intervention, and then at 12 and 24 weeks post-intervention
  * utilized to assess participant's level of perceived stress
  * 10 questions; responses from 0 to 4
  * minimum total score: 0; maximum total score: 40; higher scores indicative of higher perceived chronic levels of stress
Change in Generalized Anxiety Disorder-7 (GAD-7) scale scores | Administered prior to the intervention, and then at 12 and 24 weeks post-intervention
  * utilized in the assessment of anxiety
  * 7 questions; responses from 0 to 3
  * minimum total score: 0; maximum total score 21; higher scores indicative of severe anxiety symptoms
Change in Subjective Happiness Scale (SHS) scores | Administered prior to the intervention, and then at 12 and 24 weeks post-intervention
  * utilized to assess participant's level of global subjective happiness
  * 4 questions; responses from 1 to 7
  * minimum total score: 4; maximum total score 28; higher scores indicative of higher levels of subjective happiness

CONTACTS AND LOCATIONS:
Overall Officials: Edward Spilg, MD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Mak WW, Ng IS, Wong CC. Resilience: enhancing well-being through the positive cognitive triad. J Couns Psychol. 2011 Oct;58(4):610-7. doi: 10.1037/a0025195. PMID 21895357
- [Background] Mealer M, Jones J, Newman J, McFann KK, Rothbaum B, Moss M. The presence of resilience is associated with a healthier psychological profile in intensive care unit (ICU) nurses: results of a national survey. Int J Nurs Stud. 2012 Mar;49(3):292-9. doi: 10.1016/j.ijnurstu.2011.09.015. Epub 2011 Oct 5. PMID 21974793
- [Background] McGarry S, Girdler S, McDonald A, Valentine J, Lee SL, Blair E, Wood F, Elliott C. Paediatric health-care professionals: relationships between psychological distress, resilience and coping skills. J Paediatr Child Health. 2013 Sep;49(9):725-32. doi: 10.1111/jpc.12260. Epub 2013 Jul 1. PMID 23808920
- [Background] Lü W, Wang Z, Liu Y, Zhang H. Resilience as a mediator between extraversion, neuroticism and happiness, PA and NA. Personal Individ Differ. 2014;63:128-133
- [Background] Fox S, Lydon S, Byrne D, Madden C, Connolly F, O'Connor P. A systematic review of interventions to foster physician resilience. Postgrad Med J. 2018 Mar;94(1109):162-170. doi: 10.1136/postgradmedj-2017-135212. Epub 2017 Oct 10. PMID 29018095
- [Background] Sood A, Sharma V, Schroeder DR, Gorman B. Stress Management and Resiliency Training (SMART) program among Department of Radiology faculty: a pilot randomized clinical trial. Explore (NY). 2014 Nov-Dec;10(6):358-63. doi: 10.1016/j.explore.2014.08.002. Epub 2014 Aug 21. PMID 25443423
- [Background] Charmaz K. Constructing Grounded Theory. Sage; 2014. https://us.sagepub.com/en-us/nam/constructing-grounded-theory/book235960. Accessed December 21, 2017
- [Derived] Spilg EG, Kuk H, Ananny L, McNeill K, LeBlanc V, Bauer BA, Sood A, Wells PS. The impact of Stress Management and Resilience Training (SMART) on academic physicians during the implementation of a new Health Information System: An exploratory randomized controlled trial. PLoS One. 2022 Apr 22;17(4):e0267240. doi: 10.1371/journal.pone.0267240. eCollection 2022. Erratum In: PLoS One. 2024 Apr 11;19(4):e0302288. doi: 10.1371/journal.pone.0302288. PMID 35452478